CLINICAL TRIAL: NCT01440504
Title: Ex Vivo Evaluation of the Interest of the Association of Platinum With a Molecule BH3-mimetic ABT-737 in Samples of Ovarian Tumors
Acronym: ABT737 exvivo
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Collaborators: GRECAN (Unknown)
Responsible Party: Sponsor
Other Study IDs: ABT-737 ex vivo
Record Dates: First submitted 2011-09-15; First posted 2011-09-26 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cancer
Keywords: Cancer; Ovarian; chemotherapy; BH3-mimetic; platin; ex-vivo
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: culture ex vivo with exposure to different therapeutic agents alone or in combination. — When tumor resection, tumor specimens of ovarian cancer will be made towards a culture ex vivo with exposure to different therapeutic agents alone or in combination.

SUMMARY:
The aim of the study is to quantify the ex vivo induction of apoptosis by ABT-737 + association platinum in samples exposed and demonstrate the value of this combination compared to the agents used alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Ovarian cancer patients with at least five tumor samples does not affect the diagnosis, based on other tumor masses
* Surgery of any initial chemotherapy naive
* Patient information and signed informed consent

Exclusion Criteria:

* A person deprived of liberty or under guardianship
* Insufficient tumor samples of ovarian cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient, any chemotherapy naive or ovarian surgery, ovarian cancer with at least five tumor samples does not affect the diagnostic
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
rate of apoptotic cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: JOLY Florence, Pr, Principal Investigator — Centre françois Baclesse
Locations (1):
- Centre François Baclesse, Caen, France